CLINICAL TRIAL: NCT00515281
Title: Inhaled Nitric Oxide and Neuroprotection in Premature Infants
Acronym: NOVA2
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: The pace of patient enrolledment forced recruitment to stop after 273 patients.
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 15405A
Record Dates: First submitted 2007-08-09; First posted 2007-08-13 (Estimated); Results first posted 2024-10-17 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2024-07

CONDITIONS: Prematurity; Bronchopulmonary Dysplasia; Intraventricular Hemorrhage; Periventricular Leukomalacia
Keywords: prematurity; nitric oxide; bronchopulmonary dysplasia; intraventricular hemorrhage; periventricular leukomalacia; neurodevelopment
MeSH Terms: conditions — Premature Birth; Bronchopulmonary Dysplasia; Leukomalacia, Periventricular | interventions — Oxygen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- INO Control (Short iNO) (Placebo Comparator): INO will be given to infants in the control group for the first 7 days of the study gas, then O2 or room air, as clinically appropriate, on the 8th day, until 33 weeks corrected age
  Interventions: Drug: inhaled nitric oxide
- INO Treatment (Long iNO) (Experimental): The treatment group will receive iNO, combined with O2 or room air, until 33 weeks corrected age.
  Interventions: Drug: inhaled nitric oxide; Drug: oxygen

INTERVENTIONS:
Drug: inhaled nitric oxide — The amount of gas will be carefully controlled and adjusted to the level that best improves the function of subject's lungs. The subject will remain on inhaled nitric oxide until he/she reaches 33 weeks of gestation if assigned to the treatment arm, or until the 8th day of the study if he/she is assigned to the control arm.
  Other Names: INO
Drug: oxygen — The amount of gas will be carefully controlled and adjusted to the level that best improves the function of the subject's lungs. Subjects in the control arm of the study will receive oxygen beginning on the 8th day of the study until he/she reaches 33 weeks of gestation.
  Other Names: O2
  Arms: INO Treatment (Long iNO)

SUMMARY:
The purpose of this study is to determine whether inhaled nitric oxide improves the neurological outcome for premature infants.

DETAILED DESCRIPTION:
With the advances in modern neonatal intensive care medicine in the last 20 years, survival of extremely preterm infants weighing less than 1500g (< 3 lbs, 5 oz) has risen markedly. However, with this increased survival has come a marked increase in the number of infants with serious neurodevelopmental disabilities: Premature infants with birth weights less than 1500g who survive to go home are at significant risk for serious neurodevelopmental problems: cognitive and motor delays, blindness, deafness, and cerebral palsy. In a recent randomized, placebo-controlled clinical trial, we assessed whether giving mechanically ventilated preterm infants inhaled nitric oxide gas (iNO) for 1 week after birth decreased the incidence of death and chronic lung disease. An unanticipated outcome of that study (Schreiber et. al. 2003) and a subsequent study of those infants at 2 years of age (Mestan et. al. 2005) was that premature infants treated with inhaled nitric oxide (iNO) have improved neurodevelopmental outcomes and physical growth at 2 years corrected age, compared with placebo-treated infants (Mestan et. al. 2005). INO therapy, therefore, appears to be a new treatment to protect the premature brain during development outside the womb. The overall goal of this application is understand the efficacy of iNO treatment in improving neurodevelopmental outcomes in at-risk premature infants.

ELIGIBILITY:
Inclusion Criteria:

* Prematurity (birthweight ≤ 1500g, < 31 weeks gestation)
* Requiring respiratory support
* Admitted to the NICU at the University of Chicago

Exclusion Criteria:

* Severe congenital anomalies
* Genetic syndromes
* Extremely sick preterm infants requiring very high ventilatory pressures (OI ≥ 20)
* Premature infants judged by the physician as nonviable

Ages: 2 Hours to 72 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 273 (Actual)
Dates: Start 2008-05 (Actual); Primary Completion 2023-06-07 (Actual); Study Completion 2023-11-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael D. Schreiber, M.D., Principal Investigator — University of Chicago
Locations (1):
- The University of Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Schreiber MD, Gin-Mestan K, Marks JD, Huo D, Lee G, Srisuparp P. Inhaled nitric oxide in premature infants with the respiratory distress syndrome. N Engl J Med. 2003 Nov 27;349(22):2099-107. doi: 10.1056/NEJMoa031154. PMID 14645637
- [Background] Mestan KK, Marks JD, Hecox K, Huo D, Schreiber MD. Neurodevelopmental outcomes of premature infants treated with inhaled nitric oxide. N Engl J Med. 2005 Jul 7;353(1):23-32. doi: 10.1056/NEJMoa043514. PMID 16000353

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | INO Control (Short iNO) | INO Treatment (Long iNO)
Started | 138 | 135
Completed | 138 | 135
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | INO Control (Short iNO) | INO Treatment (Long iNO) | Total
Number analyzed (Participants) | 138 | 135 | 273
Age, Continuous [Mean (Standard Deviation); unit: Weeks] — Gestational age
  Weeks | 27.2 (2.2) | 26.8 (2.1) | 27.0 (2.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 63 | 63 | 126
  Male | 75 | 72 | 147
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black | 99 | 91 | 190
  Non-black | 39 | 44 | 83
Region of Enrollment [Number; unit: participants]
  United States | 138 | 135 | 273

OUTCOME MEASURES:

1. Primary Outcome: Neurodevelopment
Time Frame: Two years
Population: Data were not collected (due to funding cuts).
Arm/Group | INO Control (Short iNO) | INO Treatment (Long iNO)
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Bronchopulmonary Dysplasia (BPD) or Death
Description: Need for respiratory support at 36 weeks post-menstrual age, either as positive pressure or supplemental oxygen to maintain oxygen saturations >90%, or death before discharge
Time Frame: 36 weeks of age corrected (BPD) or before discharge (death)
Measure: Count of Participants; unit: Participants
Arm/Group | INO Control (Short iNO) | INO Treatment (Long iNO)
Number analyzed (Participants) | 138 | 135
Participants | 65 | 83
Statistical Analysis 1: Comparison: INO Control (Short iNO) vs INO Treatment (Long iNO); Test type: Superiority; p = 0.017, Chi-squared

3. Secondary Outcome: Death
Description: Death before discharge
Time Frame: through discharge (up to 400 days)
Measure: Count of Participants; unit: Participants
Arm/Group | INO Control (Short iNO) | INO Treatment (Long iNO)
Number analyzed (Participants) | 138 | 135
Participants | 19 | 13
Statistical Analysis 1: Comparison: INO Control (Short iNO) vs INO Treatment (Long iNO); Test type: Superiority; p = 0.288, Chi-squared

4. Secondary Outcome: Bronchopulmonary Dysplasia
Description: Need for respiratory support at 36 weeks post-menstrual age (PMA), either as positive pressure or supplemental oxygen to maintain oxygen saturations >90%
Time Frame: 36 weeks of age corrected
Measure: Count of Participants; unit: Participants
Arm/Group | INO Control (Short iNO) | INO Treatment (Long iNO)
Number analyzed (Participants) | 138 | 135
Participants | 51 | 71
Statistical Analysis 1: Comparison: INO Control (Short iNO) vs INO Treatment (Long iNO); Test type: Superiority; p = 0.009, Chi-squared

5. Secondary Outcome: Supplemental Oxygen Use
Time Frame: 40 weeks PMA
Measure: Count of Participants; unit: Participants
Arm/Group | INO Control (Short iNO) | INO Treatment (Long iNO)
Number analyzed (Participants) | 138 | 135
Participants | 30 | 28
Statistical Analysis 1: Comparison: INO Control (Short iNO) vs INO Treatment (Long iNO); Test type: Superiority; p = 0.97, Chi-squared

6. Secondary Outcome: BPD or Death in Infants Weighing < 750g
Description: Need for respiratory support at 36 weeks post-menstrual age, either as positive pressure or supplemental oxygen to maintain oxygen saturations >90%, or death before discharge among infants < 750g
Time Frame: 36 weeks of age corrected (BPD) or before discharge (death)
Measure: Count of Participants; unit: Participants
Arm/Group | INO Control (Short iNO) | INO Treatment (Long iNO)
Number analyzed (Participants) | 41 | 41
Participants | 36 | 37
Statistical Analysis 1: Comparison: INO Control (Short iNO) vs INO Treatment (Long iNO); Test type: Superiority; p = 0.72, Chi-squared

7. Secondary Outcome: BPD or Death in Infants Weighing 750-999g
Description: Need for respiratory support at 36 weeks post-menstrual age, either as positive pressure or supplemental oxygen to maintain oxygen saturations >90%, or death before discharge among infants 750-999g
Time Frame: 36 weeks of age corrected (BPD) or before discharge (death)
Measure: Count of Participants; unit: Participants
Arm/Group | INO Control (Short iNO) | INO Treatment (Long iNO)
Number analyzed (Participants) | 43 | 44
Participants | 20 | 36
Statistical Analysis 1: Comparison: INO Control (Short iNO) vs INO Treatment (Long iNO); Test type: Superiority; p < 0.001, Chi-squared

8. Secondary Outcome: BPD or Death in Black Infants
Description: Need for respiratory support at 36 weeks post-menstrual age, either as positive pressure or supplemental oxygen to maintain oxygen saturations >90%, or death before discharge among Black infants
Time Frame: 36 weeks of age corrected (BPD) or before discharge (death)
Measure: Count of Participants; unit: Participants
Arm/Group | INO Control (Short iNO) | INO Treatment (Long iNO)
Number analyzed (Participants) | 99 | 91
Participants | 50 | 53
Statistical Analysis 1: Comparison: INO Control (Short iNO) vs INO Treatment (Long iNO); Test type: Superiority; p = 0.28, Chi-squared

ADVERSE EVENTS:
Time Frame: through discharge (up to 400 days)
Description: Standard perinatal morbidities were tracked and reported and all are considered serious adverse events (SAEs). Non-serious adverse events were not defined or tracked.
Arm/Group | INO Control (Short iNO) | INO Treatment (Long iNO)
All-Cause Mortality (participants affected / at risk) | 19/138 | 13/135
Serious Adverse Events (participants affected / at risk) | 53/138 | 61/135
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | INO Control (Short iNO) (N=138) | INO Treatment (Long iNO) (N=135)
Severe IVH/PVL (Vascular disorders) | 13 | 16 — Severe intraventricular hemorrhage (IVH) or periventricular leukomalacia (PVL)
Pulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 2 | 5 — Acute bleeding from the lung, from the upper respiratory tract and the trachea, and the pulmonary alveoli.
Pneumorthorax (Respiratory, thoracic and mediastinal disorders) | 13 | 10 — Collapsed lung
Pulmonary interstitial emphysema (PIE) (Respiratory, thoracic and mediastinal disorders) | 19 | 26 — A condition where air dissects through alveolar walls into the adjacent interstitial tissues where it forms cystic spaces with an associated inflammatory reaction.
Symptomatic patent ductus arteriosis (PDA) (Cardiac disorders) | 45 | 41 — An opening between the two main vessels leading to the heart
Necrotizing enterocolitis (NEC) of Bell's stage 2 severity or greater (Gastrointestinal disorders) | 14 | 19 — Inflammatory disease of the newborn bowel.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2017-05-10): https://cdn.clinicaltrials.gov/large-docs/81/NCT00515281/Prot_SAP_ICF_000.pdf